CLINICAL TRIAL: NCT05485012
Title: Modulation of Drug Intake: Evaluation of Opioid and Cannabinoid Interactions on Drug Self-Administration
Brief Title: Reinforcing Effects of Marijuana and Opioids
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanna Babalonis, PhD (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Shanna Babalonis, PhD, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 45017-20221; R01DA045700 (NIH)
Record Dates: First submitted 2022-07-18; First posted 2022-08-02 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Marijuana Use; Opioid Use
Keywords: marijuana; opioid; healthy participants; laboratory study
MeSH Terms: conditions — Marijuana Use; Marijuana Abuse | interventions — nabiximols; Analgesics, Opioid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Double-blind marijuana/placebo administration (Experimental): Participants will receive double-blind administration of vaporized marijuana/placebo
  Interventions: Drug: Marijuana; Drug: Opioid
- Double-blind opioid/placebo administration (Experimental): Participants will receive double-blind administration of intranasal opioid agonist/placebo
  Interventions: Drug: Marijuana; Drug: Opioid

INTERVENTIONS:
Drug: Marijuana — Double-blind administration of marijuana
  Other Names: Cannabis
Drug: Opioid — Double-blind administration of an opioid agonist

SUMMARY:
The primary goals of this study are to examine 1) marijuana modulation of oxycodone self-administration and 2) oxycodone modulation of marijuana self-administration, under controlled conditions and across a range of doses for each drug.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-50
* Experience with marijuana and opioids
* General good health
* Willing to live at the University of Kentucky Hospital (research unit) for approx. 6.5 weeks (meals are provided,

Exclusion Criteria:

* Significant medical complications/conditions

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2023-08-03 (Actual); Primary Completion 2025-03-27 (Actual); Study Completion 2025-03-27 (Actual)

PRIMARY OUTCOMES:
Self-Administration | Collected once during each self-administration session
  The number of units of drug earned in each session

SECONDARY OUTCOMES:
Subjective measures | Baseline, post-dose during each session (change from baseline is assessed); visual analog scales will be the primary measure (0-100, 0=not at all, 100=extremely)
  Ratings of drug effects (e.g., feeling high, impaired, good drug effects)
Heart rate | Baseline, post-dose during each session (change from baseline is assessed)
  Beats per minute
Blood pressure | Baseline, post-dose during each session (change from baseline is assessed)
  Systolic and diastolic blood pressure (mm/hg)

CONTACTS AND LOCATIONS:
Overall Officials: Shanna Babalonis, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-03-12): https://cdn.clinicaltrials.gov/large-docs/12/NCT05485012/ICF_000.pdf